CLINICAL TRIAL: NCT02805842
Title: Evaluation of Incidence of Non Adherence to Treatment With Once-daily Formulation of Tacrolimus (ADVAGRAF) in Kidney Transplant Recipients
Brief Title: Incidence of Non Adherence to Treatment With Once-daily Formulation of Tacrolimus
Acronym: Advagraf
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry); Teva Pharma (Industry)
Responsible Party: Principal Investigator, Alexander yussim, Director transplantation research unit, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0076-16 RMC
Record Dates: First submitted 2016-05-08; First posted 2016-06-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Medication Adherence
Keywords: non adherence; Tacrolimus; Advagraf
MeSH Terms: conditions — Medication Adherence | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus BID (Active Comparator): 20 patients receiving twice daily (BID) Tacrolimus
  Interventions: Drug: Tacrolimus BID
- Advagraf QD (Active Comparator): 40 patients randomized to receive once daily (QD) Advagraf
  Interventions: Drug: Advagraf QD

INTERVENTIONS:
Drug: Tacrolimus BID — Administration of Tacrolimus BID
  Other Names: Prograf, Tacrocell
  Arms: Tacrolimus BID
Drug: Advagraf QD — administration of Advagraf QD
  Other Names: Advagraf
  Arms: Advagraf QD

SUMMARY:
Aim The primary objective of this study is to compare medication adherence with medical therapy in patients receiving once-daily versus twice-daily tacrolimus regimens.

Participants 60 adult renal transplant patients randomized 1:2 into twice-daily and once-daily tacrolimus groups

Outcomes The primary outcome will be medication adherence to the once-daily and twice-daily regimens, measured in terms of implementation. Secondary outcomes will include graft and patient survival, renal function and adverse events. Follow up - 12 months

DETAILED DESCRIPTION:
Following randomization (Day 0), 60 kidney transplant recipients of deceased or live kidneys will be randomized 1:2 into control and study- experimental arm. In control arm, named Tacrolimus BID arm, tacrolimus will be administered unchanged twice daily, morning and evening, while in study--experimental group named Tacrolimus QD- Advagraf, the Advagraf tacrolimus formulation will be administered once daily in the morning. In both groups doses will be adjusted to maintain tacrolimus trough levels at 10-12 ng/mL (days 1-28), 8-10 ng/mL (days 29-168) and 6-8 ng/mL thereafter for both treatment arms.

Adjunct immunosuppression. Per-protocol rejection prophylaxis: All patients will receive Basiliximab induction at 20mg/bw on days 0 and 4. Methylprednisolone will be administered as intravenous bolus doses of 500 mg , 250 mg and 125 mg perioperatively, on days 0,1 and 2. Thereafter oral prednisone will be given: 20 mg/day (days 2-14), 15 mg/day (days 15-30), 10 mg/day (days 30-45), 7.5 mg/day (days 45-60) and 5 mg/day thereafter. MMF (2 g BID) will be started preoperatively, and reduced to 500 mg three times daily after 14-30 days.

Rejection treatment: First-line acute rejection (AR) therapy with corticosteroids will be administered at the dose of 500 mg/day for 3 days. Mono- and/or polyclonal antibodies could be used as therapy for corticosteroid-resistant AR. First-line antibody therapy will be permitted only if biopsy indicate a severe vascular rejection (Banff IIB or III).

Prophylactic treatment:

Prophylactic antiviral treatment with oral ganciclovir 450 mg/day, and PCP prevention with 400 mg Sulfamethoxazole and 80 mg of Trimethoprim/day will be given to all patients on days 1-90.

Endpoints.

The primary endpoint:

• adherence to the Tacrolimus administration defined as self-reported number of missed drug ingestions scored in Morisky Medical Adherence Assessment questionnaire

Secondary endpoints:

• efficacy failure defined as biopsy proven rejection, renal function, incidence of adverse events (AEs) and graft loss or death at the end of the analysis period

Statistical analysis The data collected will be analyzed with Fisher's exact test, Wilcoxon' matched pair test and Kaplan-Meier's test

ELIGIBILITY:
Inclusion Criteria

* Age: 18 Years to 60 Years
* Gender: both
* Patients willing and able to participate in this study
* Patients who signed the informed consent form
* Patients who can visit the center based on the study schedule in the protocol

Exclusion Criteria

* Patients who had previously received a kidney or another organ
* Patients, having positive lymphocyte cross-match
* Patients with PRA >50%
* Patients, who underwent desensitization
* Patients, who were diagnosed with cancer in the last five years
* Patients, who themselves or their donors have positive HIV, HBsAg, or anti-HCV test results
* Patients, who were treated with other investigated drugs within 30 days from their study enrollment
* Patients, who are planning to be pregnant, or who are pregnant or breastfeeding and who are not planning to use any contraceptive method during the study period.
* Patients who were addicted to drugs/alcohol within six months of their study enrollment
* Patients, who have a mental illness that makes appropriate communication with them impossible

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Morisky Medical Adherence Assessment questionnaire | 2 years
  adherence to the Tacrolimus QD administration defined as self-reported number 9on scale from 1-8) of missed drug ingestions scored in Morisky Medical Adherence Assessment questionnaire

SECONDARY OUTCOMES:
graft and patient survival | 2 years
  % of patients and grafts alive after 1st and 2nd year of study
gfr | 2 years
  gfr - glomerular filtration rate - a measure of renal function, in ml/min/1.73m2
adverse events | 2years
  percentage of patients with complications

CONTACTS AND LOCATIONS:
Overall Officials: Eyan Mor, MD, Study Director — Rabin Med CTR
Locations (1):
- Rabin Med Ctr, Petah Tikva, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829